CLINICAL TRIAL: NCT06232746
Title: Creation of Side-to-Side Compression Anastomosis Using the GT Metabolic Solutions DI Biofragmentable Magnetic Anastomosis System (Magnet System, DI Biofragmentable) to Achieve Jejuno-Ileal Diversion in Adults With Obesity and Type 2 Diabetes Mellitus: MJI Study
Brief Title: Magnetic Jejuno-Ileal Diversion Study ("MJI Study")
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GT Metabolic Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTM-008
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is an open-label single-center study enrolling up to 10 subjects in the Czech Republic
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnet System, DI Biofragmentable (Experimental): GT Metabolic Solutions DI Biofragmentable Magnetic Anastomosis System (Magnet System, DI Biofragmentable)
  Interventions: Device: Magnet System, DI Biofragmentable

INTERVENTIONS:
Device: Magnet System, DI Biofragmentable — Anastomoses achieved by magnetic compression.

SUMMARY:
The purpose of this clinical research study is to evaluate the feasibility/performance, safety and initial efficacy of the GT Metabolic Solutions DI Biofragmentable Magnetic Anastomosis System (Magnet System, DI Biofragmentable and hereafter referred to as the DI Magnet System) for creation of a side-to-side jejuno-ileal anastomosis in adults with obesity and type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
The purpose of this clinical research study is to evaluate the feasibility/performance, safety and initial efficacy of the GT Metabolic Solutions DI Biofragmentable Magnetic Anastomosis System (Magnet System, DI Biofragmentable and hereafter referred to as the DI Magnet System) for creation of a side-to-side jejuno-ileal anastomosis in adults with obesity and type 2 diabetes mellitus (T2DM). This partial diversion of intestinal contents from jejunum to the ileum is intended to facilitate weight management/loss and improve metabolic outcomes. Side-by side anastomoses are currently created by sutures, staples, and anastomotic compression devices. This study explores a partial jejuno-ileal diversion procedure creating a side-to-side anastomosis with magnetic compression anastomosis.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age, inclusive, at the time of informed consent
2. BMI 30-40 kg/m2
3. T2DM (defined as HbA1c ≥ 6.5%) without previous sleeve gastrectomy and without plan to perform a concurrent sleeve gastrectomy
4. Agrees to refrain from any type of additional bariatric or reconstructive surgery that would affect body weight for the duration of the study
5. If a child-bearing female, subject must commit to not becoming pregnant and agree to use contraception for the duration of the study
6. Willing and able to comply with protocol requirements

Exclusion Criteria:

1. Type 1 diabetes
2. Use of injectable insulin
3. Uncontrolled T2DM
4. Plan to perform a sleeve gastrectomy with the jejuno-ileal anastomosis procedure
5. Uncontrolled hypertension, dyslipidemia or sleep apnea
6. Prior intestinal, colonic or duodenal surgery, other than bariatric
7. Prior surgery, trauma, prostheses, disease or genetic expression which prevent or contra-indicate the procedure, including scarring and abnormal anatomy.
8. Refractory gastro-esophageal reflux disease (GERD)
9. Barrett's disease
10. Helicobacter pylori positive and/or active ulcer disease
11. Large hiatal hernia
12. Inflammatory bowel or colonic diverticulitis disease
13. Any anomaly precluding orogastric access by gastroscope and catheters, and manipulation techniques.
14. Implantable pacemaker or defibrillator
15. Psychiatric disorder, except well-controlled depression with medication for > 6 months
16. History of substance abuse
17. Woman who is either pregnant or breast feeding
18. Woman of childbearing potential who does not agree to use an effective method of contraception.
19. Any comorbidity or current status of subject's physiological fitness that in the surgeon's or anesthesiologist's opinion represents safety concerns that make the subject medically unfit for the procedure, including any significant congenital or acquired anomalies of the GI tract at or distal to the placement of the magnets.
20. Unhealed ulcers, bleeding lesions, tumor, or any other lesion at target magnet deployment site
21. Expected need for MR imaging within the first 2 months after the procedure
22. Any anomaly preventing/contraindicating endoscopic or laparoscopic access and procedures
23. Had surgical or interventional procedure within 30 days prior to procedure
24. Any scheduled surgical or interventional procedure planned within 30 days postprocedure
25. Any stroke/TIA within 6 months prior to consent
26. Requires chronic anticoagulation therapy (except aspirin)
27. Active infections requiring antibiotic therapy, unless resolved before undergoing the study procedure
28. Unable to comply with the follow-up schedule and assessments
29. Recent tobacco or nicotine product cessation within < 3 months prior to informed consent
30. Known allergies to the device components or contrast media
31. Limited life expectancy due to terminal disease
32. Currently participating in another clinical research study with an investigational drug or medical device
33. Any condition that, in the investigator's opinion, may preclude completion of followup assessments through Day 360 (e.g., a medical condition that may increase the risk associated with study participation or may interfere with interpretation of study results, inability to adhere to the visit schedule, or poor compliance with treatment regimen)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Feasibility and performance of the side-to-side anastomosis for jejuno-ileal diversion using the DI Magnet System. | From date of study index procedure through 90 days
  The jejuno-ileal diversion will be considered feasible if it results in successful:
  * Placement of the Magnet System (≥ 90% alignment of magnets); and
  * Creation of a patent anastomosis confirmed radiologically, and
  * Passage of magnets without any surgical re-interventions.
  The primary endpoint will be met if the feasibility/performance is confirmed in ≥ 80% of enrolled and treated participants.
Safety of the DI Magnet System | Procedure, Day 90, Day 180, Day 360
  Freedom from serious adverse events related to the study device or study device procedure requiring additional emergency surgery or re-intervention, including:
  * All-cause mortality
  * Intestinal perforation and/or peritonitis
  * Intestinal obstruction
  * Life-threatening bleeding
  * Incidence of device malfunctions

CONTACTS AND LOCATIONS:
Locations (1):
- OB KLINIKA a.s., Prague, Czechia

IPD SHARING:
Plan to Share IPD: No